CLINICAL TRIAL: NCT05259033
Title: A 52 Week Study Comparing the Efficacy and Safety of Once Weekly IcoSema and Once Weekly Semaglutide, Both Treatment Arms With or Without Oral Anti Diabetic Drugs, in Participants With Type 2 Diabetes Inadequately Controlled With a GLP 1 Receptor Agonist. COMBINE 2
Brief Title: A Research Study to See How Well the New Weekly Medicine IcoSema, Which is a Combination of Insulin Icodec and Semaglutide, Controls Blood Sugar Level in People With Type 2 Diabetes Compared to Weekly Semaglutide (COMBINE 2)
Acronym: COMBINE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1535-4592; U1111 1260 8268 (Other: World Health Organization (WHO)); 2020 005308 21 (EudraCT Number)
Record Dates: First submitted 2022-02-10; First posted 2022-02-28 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IcoSema (Experimental): Participants will get once weekly dose
  Interventions: Drug: IcoSema
- Semaglutide (Experimental): Participants will get once weekly dose
  Interventions: Drug: Semaglutide 1 mg

INTERVENTIONS:
Drug: IcoSema — IcoSema once weekly subcutaneously (s.c., under the skin) using a needle and a pen.
  For about 1 year and 1 month.
  Arms: IcoSema
Drug: Semaglutide 1 mg — Semaglutide once weekly subcutaneously (s.c., under the skin). Dose titrated to 1mg over 8 weeks (0.25 mg for 4 weeks, 0.5 mg for 4 weeks). For about 1 year and 1 month.
  Arms: Semaglutide

SUMMARY:
This study will compare the new medicine IcoSema, which is a combination of insulin icodec and semaglutide, taken once a week, to semaglutide taken once a week in people with type 2 diabetes.

The study will look at how well IcoSema controls blood sugar level in people with type 2 diabetes compared to semaglutide.

Participants will either get IcoSema or semaglutide. Which treatment participants get is decided by chance. IcoSema is a new medicine that doctors cannot prescribe. Doctors can already prescribe semaglutide in many countries.

Participants will get IcoSema or semaglutide, which they must inject once a week with a pen, which has a small needle, in a skin fold in the thigh, upper arm, or stomach.

The study will last for about 1 year and 1 month. Participants will have 18 clinic visits, 34 phone/video calls with the study doctor, and 4 contacts with the site that can either be clinic visits or phone/video calls.

At 11 clinic visits participants will have blood samples taken. At 7 clinic visits participants cannot eat or drink (except for water) for 8 hours before the visit.

Women cannot take part if pregnant, breast-feeding or plan to get pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with type 2 diabetes mellitus 180 days or more before screening.
* HbA1c of 7.0 - 10.0% (53.0 - 85.8 mmol/mol) (both inclusive) as assessed by central laboratory on the day of screening.
* Insulin naïve. The following exceptions are permitted: short term insulin treatment for a maximum of 14 days before screening and/or prior insulin treatment for gestational diabetes.
* Treated with stable doses of daily or weekly GLP-1 receptor agonist (excluding once weekly semaglutide with doses higher than 1.0 mg) according to local label for the treatment of diabetes for 90 days or more before screening. The treatment can be with or without any of the following anti diabetic drugs with stable doses for 90 days or more before screening: Metformin - Sulfonylureas (Sulfonylureas, meglitinides (glinides) and DPP 4 inhibitors must be discontinued at randomisation) - Meglitinides (glinides)(Sulfonylureas, meglitinides (glinides) and DPP 4 inhibitors must be discontinued at randomisation) - DPP 4 inhibitors (Sulfonylureas, meglitinides (glinides) and DPP 4 inhibitors must be discontinued at randomisation) - Sodium glucose co transporter 2 inhibitors - Alpha-glucosidase inhibitors - Thiazolidinediones - Marketed oral combination products only including the products listed above.
* Body mass index (BMI) below or equal to 40.0 kg/m^2.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Anticipated initiation or change in concomitant medication (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or systemic corticosteroids).
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening.
* Any episodes (as declared by the participant or in the medical records) of diabetic ketoacidosis within 90 days before screening.
* Presence or history of pancreatitis (acute or chronic) within 180 days before screening.
* Any of the following: Myocardial infarction, stroke, hospitalization for unstable angina pectoris or transient ischaemic attack within 180 days before screening.
* Chronic heart failure classified as being in New York Heart Association Class IV at screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days before screening or in the period between screening and randomisation. Pharmacological pupil dilation is a requirement unless using a digital fundus photography camera specified for non dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 683 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (135):
- United States (50):
  - Univ of AL at Birmingham_BRM, Birmingham, Alabama
  - Pri Med Grp dba/Gil Ctr Fam, Gilbert, Arizona
  - Clinical Research Institute of Arizona, Sun City West, Arizona
  - John Muir Physicians Network, Concord, California
  - Velocity Clin Res Los Angeles, Los Angeles, California
  - Velocity Clin Res Wstlke, Los Angeles, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Premier Medical Center, Inc., Toluca Lake, California
  - Northeast Research Institute, Fleming Island, Florida
  - Northeast Res Inst. Inc., Jacksonville, Florida
  - Est Cst Inst for Rsrch,Jksnvil, Jacksonville, Florida
  - South Broward Research LLC, Miramar, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Florida Institute For Clinical Research, Orlando, Florida
  - Oviedo Medical Research, LLC, Oviedo, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Javara/Privia Med Grp GA,LLC, Albany, Georgia
  - East West Med Res Inst, Honolulu, Hawaii
  - Saltzer Medical Group Research, Nampa, Idaho
  - Endeavor Health, Skokie, Illinois
  - Ileana J Tandron APMC, Slidell, Louisiana
  - MedStar Hlth Res Institute, Hyattsville, Maryland
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - John J Shelmet, MD, Lawrenceville, New Jersey
  - Albuquerque Clin Trials, Inc., Albuquerque, New Mexico
  - Southgate Medical Group, LLP, West Seneca, New York
  - PharmQuest Life Sciences LLC, Greensboro, North Carolina
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - Thomas Jefferson Univ Di Rsrch Ctr, Philadelphia, Pennsylvania
  - Palmetto Clinical Research, Summerville, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - Diabetes and Thyroid Ctr of FW, Fort Worth, Texas
  - DCOL Ctr for Clin Res, Longview, Texas
  - Texas Diabetes & Endocrinology_Round Rock, Round Rock, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Sugar Lakes Family Practice PA, Sugar Land, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Javara Inc. / Privia Medical Group LLC_Forest, Forest, Virginia
  - Javara Inc/Privia Md GpLLC Fst, Forest, Virginia
  - TPMG Clinical Research, Newport News, Virginia
- Brazil (6):
  - Centro de Diabetes Metabolismo e Endocrinologia, Fortaleza, Ceará
  - Instituto de Ciências Farmacêuticas de Estudos e Pesquisas, Aparecida de Goiânia, Goiás
  - Quanta Diagnóstico Nuclear / Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - BR Trials - Ensaios Clínicos e Consultoria Ltda., São Paulo, São Paulo
- Canada (10):
  - LMC Clinical Res Thornhill, Concord, Ontario
  - Medical Trust Clinics, Inc., Courtice, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Western Univ. Cnt for Studies in Fam Med, London, Ontario
  - Bluewater Clin Res Group,Inc, Sarnia, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - Recherche GCP Research, Montreal, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Montreal, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
  - Recherche Clinique Sigma inc, Québec
- China (12):
  - Anhui Provincial Hospital-Endocrinology, Hefei, Anhui
  - Peking University People's Hospital-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Huizhou Central People's Hospital-Endocrinology, Huizhou, Guangdong
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - Jinan Central Hospital, Ji'nan, Shandong
  - Huashan Hospital Fudan University-Endocrinology, Shanghai, Shanghai Municipality
  - Shanghai Huashan Hospital, Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality
  - Tianjin Medical University Chu Hsien-I Memorial Hospital-Endocrinology, Tianjin, Tianjin Municipality
- France (6):
  - Centre Hospitalier Universitaire de Rouen - Hopital de Bois Guillaume, Bois-Guillaume
  - Les Hopitaux de Chartres-Hopital Louis Pasteur, Le Coudray
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-1, Le Creusot
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-2, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Greece (8):
  - Evangelismos Hospital, Athens
  - Iatriko Psychicou Private Clinic, Athens
  - 'G. Gennimatas' General Hospital of Athens, Athens
  - Univ Gen Hospital Larisa, Larissa
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
- Hungary (4):
  - PTE-AOK II. Belgyogyaszati Klinika es Nephrologiai Centrum, Pécs, Baranya Vármegye
  - Debreceni Egyetem Belgyógyászati Klinika, Debrecen, Hajdú-Bihar
  - Debreceni Egyetem Klinikai Központ Belgyógyászati Klinika D épület, Debrecen, Hajdú-Bihar
  - MED-TIMA Kft., Budapest
- Israel (6):
  - Clalit sick fund Herzeliya, Herzeliya, Israel
  - Linn clinic - Clalit Health Services, Haifa
  - Diabetes Clinic Wolfson MC, Holon
  - Diabetes Unit Hadassah Ein Karem MC, Jerusalem
  - Diabetes Clinic Meir MC, Kfar Saba
  - Endrocrinolgy Clinic - Sheba Medical Center, Tel Litwinsky
- Japan (9):
  - Heiwadai Hospital, Miyazaki, Miyazaki
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Futata Tetsuhiro Clinic Meinohama, Fukuoka-shi, Fukuoka
  - Gifu University Hospital, Gifu
  - Naka Kinen Clinic, Ibaraki
  - Takatsuki Red Cross Hospital, Osaka
  - Shimizu Clinic Fusa, Saitama
  - Soka Sugiura Internal Medicine Clinic_Internal Medicine, Saitama
  - Shinden Higashi Clinic, Sendai-shi, Miyagi
- Russia (7):
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - National Medical Research Center of Endocrinology, Moscow
  - Limited Law Company "Healthy Family" Medicine Center", Novosibirsk
  - BHI of Omsk Region "City Hospital № 3", Omsk
  - Penza Regional Clinical Hospital named after N.N. Burdenko, Penza
  - Rostov State Medical University_Rostov-on-Don, Rostov-on-Don
  - Polyclinic #2 in Yoshkar-Ola, Yoshkar-Ola
- Slovakia (6):
  - DIOLI s.r.o., Košice
  - HUMAN-CARE s.r.o., Košice
  - DIADAN, s.r.o. Kosice, Košice
  - FNsP L. Pasteura, Košice
  - DIA - KONTROL s.r.o., Levice
  - MUDr. Alena Lomencikova, s.r.o, Turčianske Teplice
- Sweden (3):
  - Primary Care Trial Center, PTC ,Gothia Forum, Gothenburg
  - Enheten för Kliniska Studier (EKS), Örebro, Örebro
  - Centrum for Diabetes, Academical Specialist Centrum, Stockholm
- Switzerland (3):
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital Olten, Olten
  - Diabetes Adipositas Zentrum Zürich, Zollikerberg
- Taiwan (5):
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Lingvay I, Benamar M, Chen L, Fu A, Jodar E, Nishida T, Riveline JP, Yabe D, Zueger T, Rea R. Once-weekly IcoSema versus once-weekly semaglutide in adults with type 2 diabetes: the COMBINE 2 randomised clinical trial. Diabetologia. 2025 Apr;68(4):739-751. doi: 10.1007/s00125-024-06348-5. Epub 2025 Jan 17. PMID 39820580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 124 sites in 13 countries.
Pre-assignment Details: Participants were randomised in 1:1 ratio to receive subcutaneous (s.c.) injection of either IcoSema or semaglutide once weekly. The trial had a 52-week treatment period followed by a 5-week follow-up period.
Groups:
- IcoSema: Participants received once weekly 700 units per millilitre (U/mL) of insulin icodec and 2 milligram per millilitre (mg/mL) of semaglutide subcutaneously for 52 weeks. Participants were to perform once daily pre-breakfast self-monitoring plasma glucose (SMPG). The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: < 4.4 mmol/L: dose re-duced by 10 U; 4.4-7.2 mmol/L: no adjustment; > 7.2 mmol/L: dose increased by 10 U. Dose titration of IcoSema was based on the respective premeal(s) and bedtime self-measured plasma glucose (SMPG) measured weekly.
- Semaglutide: Participants received once weekly semaglutide subcutaneously in a dose escalation manner, with dose increases every 4 weeks for up to week 8 (0.25 milligrams [mg], 0.5 mg) followed by dose of 1.0 mg once weekly up to the end of treatment period.
Period: Overall Study
Arm/Group | IcoSema | Semaglutide
Started | 342 | 341
Full Analysis Set | 342 | 341
Safety Analysis Set | 341 | 340
Treated | 341 | 340
Completed | 329 | 336
Not Completed | 13 | 5
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | IcoSema | Semaglutide | Total
Number analyzed (Participants) | 342 | 341 | 683
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (10.5) | 58.3 (9.8) | 59.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 145 | 286
  Male | 201 | 196 | 397
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 37 | 74
  Not Hispanic or Latino | 285 | 289 | 574
  Unknown or Not Reported | 20 | 15 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 99 | 90 | 189
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 9 | 21
  White | 210 | 224 | 434
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) to week 52 in HbA1c is presented.The outcome measure was evaluated based on the data from in study period, where all data from randomisation until last date of any of the following: 1) last direct participant-site contact; 2) participants who withdrew their informed consent; 3) last participant-investigator contact as defined by the investigator for participants who lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death of participants who died before any of the above.
Time Frame: Baseline (week 0), (week 52)
Population: Full Analysis Set (FAS) which comprised all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | IcoSema | Semaglutide
Number analyzed (Participants) | 325 | 335
Percentage point of HbA1c | -1.40 (0.91) | -0.86 (0.96)
Statistical Analysis 1: Comparison: IcoSema vs Semaglutide; Treatment policy strategy; Test type: Superiority — Responses were analysed using an analysis of covariance (ANCOVA) model with region and randomised treatment as fixed factors and baseline HbA1c as covariate. Each imputed dataset is analysed separately and estimates are combined using Rubin's rules; p < 0.0001, ANCOVA; Estimated treatment difference = -0.44, 95% CI 2-sided [-0.56 to -0.33]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) to week 52 in FPG is presented.The outcome measure was evaluated based on the data from in study period, where all data from randomisation until last date of any of the following: 1) last direct participant-site contact; 2) participants who withdrew their informed consent; 3) last participant-investigator contact as defined by the investigator for participants who lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death of participants who died before any of the above.
Time Frame: Baseline (week 0), (week 52)
Population: FAS which comprised all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | IcoSema | Semaglutide
Number analyzed (Participants) | 313 | 317
Millimoles per litre (mmol/L) | -2.74 (2.85) | -1.41 (2.89)

3. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline (week 0) to week 52 in body weight is presented. The outcome measure was evaluated based on the data from in study period, where all data from randomisation until last date of any of the following: 1) last direct participant-site contact; 2) participants who withdrew their informed consent; 3) last participant-investigator contact as defined by the investigator for participants who lost to follow-up (i.e. possibly an unscheduled phone visit); 4) death of participants who died before any of the above.
Time Frame: Baseline (week 0), (week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | IcoSema | Semaglutide
Number analyzed (Participants) | 325 | 336
Kilogram (kg) | 0.89 (4.36) | -3.77 (4.60)

4. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 Milligram Per Decilitre [mg/dL]) , Confirmed by Blood Glucose [BG] Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association/ International Hypoglycaemia Study Group, where glycemic criteria for level 2 was less than (<) 3.0 mmol/L (54 mg/dL) and level 3 had no specific glucose threshold. The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1)last follow-up visit (V56); 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: Week 0 to Week 57
Population: Safety Analysis Set (SAS) included all participants exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | IcoSema | Semaglutide
Number analyzed (Participants) | 341 | 340
Episodes | 15 | 13

5. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by BG Meter)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association/ International Hypoglycaemia Study Group, where glycemic criteria for level 2 was < 3.0 mmol/L (54 mg/dL). The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1)last follow-up visit (V56); 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: Week 0 to Week 57
Population: SAS included all participants exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | IcoSema | Semaglutide
Number analyzed (Participants) | 341 | 340
Episodes | 15 | 13

6. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Hypoglycaemic episodes were classified according to the American Diabetes Association/ International Hypoglycaemia Study Group, where glycemic criteria for level 3 had no specific glucose threshold.The outcome measure was evaluated based on data from on treatment period, where all data from date of first dose of randomised treatment as recorded on the electronic case report form (eCRF) until the first date of any of the following: 1)last follow-up visit (V56); 2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after the end of the dosing interval for both treatment arms); 3) end-date for the in-study data points sets.
Time Frame: Week 0 to Week 57
Population: SAS included all participants exposed to randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | IcoSema | Semaglutide
Number analyzed (Participants) | 341 | 340
Episodes | 0 | 0

ADVERSE EVENTS:
Time Frame: Week 0 to week 57
Description: Presented AEs are TEAEs, defined as event with onset during on treatment period where all data from date of first dose of randomised treatment as recorded on electronic case report form (eCRF) until first date of any of the below:1) last follow up visit;2) last date on randomised treatment +6 weeks (corresponding to 5 weeks after end of dosing interval for both arms);3) end-date for in-study data points. AEs were assessed in SAS and All-Cause Mortality was assessed for all enrolled participants.
Arm/Group | IcoSema | Semaglutide
All-Cause Mortality (participants affected / at risk) | 2/342 | 0/341
Serious Adverse Events (participants affected / at risk) | 38/341 | 21/340
Other Adverse Events (participants affected / at risk) | 163/341 | 159/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IcoSema (N=341) | Semaglutide (N=340)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1)
Colon dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Migraine without aura (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IcoSema (N=341) | Semaglutide (N=340)
COVID-19 (Infections and infestations) | 51 (52) | 49 (53)
Constipation (Gastrointestinal disorders) | 11 (14) | 17 (26)
Diabetic retinopathy (Eye disorders) | 19 (20) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 38 (53) | 41 (82)
Headache (Nervous system disorders) | 20 (25) | 6 (6)
Nasopharyngitis (Infections and infestations) | 33 (45) | 33 (45)
Nausea (Gastrointestinal disorders) | 40 (65) | 39 (73)
Upper respiratory tract infection (Infections and infestations) | 22 (34) | 29 (34)
Vomiting (Gastrointestinal disorders) | 17 (24) | 22 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT05259033/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT05259033/SAP_001.pdf